CLINICAL TRIAL: NCT02530658
Title: Genomes for Kids (G4K)
Brief Title: Next Generation Sequencing of Normal Tissues Prospectively in Pediatric Oncology Patients
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: G4K
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Solid, Liquid, Central Nervous System Tumors
Keywords: Genetic Predisposition; Pediatric; Genomic Analysis; Heritable Disease; Cancer Risk; Genetic Counseling; DNA; Clinical Genomics; Clinical Decision-Making; Treatment Planning; Germline
MeSH Terms: conditions — Central Nervous System Neoplasms; Genetic Predisposition to Disease | interventions — Demography; Surveys and Questionnaires; Interviews as Topic; Blood Specimen Collection; Phlebotomy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Normal tissue (germline) will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: St. Jude patients with a diagnosed solid or liquid tumor (benign or malignant) and their biological parents or legally authorized representative.
  Interventions: Study Introduction Visit, Informed Consent Visit, Informed Consent Follow-Up Visit, Return of Results Conversation, two Return of Results Follow-Up Visits, Tissue Sample (when available), Blood Sample or Skin Biopsy.
  Interventions: Other: Study Introduction Visit; Other: Informed Consent Visit; Other: Informed Consent Follow-Up Visit; Other: Return of Results Conversation; Other: Return of Results Follow-Up Visits; Procedure: Blood Sample; Procedure: Skin Biopsy

INTERVENTIONS:
Other: Study Introduction Visit — Within 5±3 weeks following arrival at SJCRH, or at the participant/family's convenience, participants will meet with a genetic counselor and clinician, provide information for a family pedigree, undergo a physical and discuss germline testing options. Study introduction materials will be provided. Families interested in the G4K study will be referred to the study nurse or other G4K member and an Informed consent visit will be scheduled.
Other: Informed Consent Visit — Within 1±3 weeks following the Study Introduction Visit, or at the participant/family's convenience, the research nurse or other study team member will consent the family and collect demographic and medical information. Participants will complete assessment questionnaires.
  Other Names: Demographic and Medical forms; Questionnaires
Other: Informed Consent Follow-Up Visit — At or after enrollment but before the release of the gerline results, or at the participant/family's convenience, a subset of participants (30-40) will participate in semi-structured interviews.
  Other Names: Interviews
Other: Return of Results Conversation — Participants will complete the assessment questionnaires.
  Other Names: Questionnaires; Interviews
Other: Return of Results Follow-Up Visits — Return of Results Follow-Up Visits will be conducted twice: the first within 8±4 weeks of the Return of Results Conversation, or at the participant/family's convenience, and the second within 28 ± 4 weeks of the Return of Results Conversation or at the participant/family's convenience. At each visit, participants will complete assessment questionnaires. Semi-structured interviews with parents and adolescents will be conducted.
  Other Names: Questionnaires; Interviews
Procedure: Blood Sample — For patients who have not previously provided a blood sample, a sample of blood will be obtained as a source of germline DNA.
  Other Names: Phlebotomy
Procedure: Skin Biopsy — After consent, for participants with a diagnosis where peripheral blood is likely to be contaminated by tumor cells, skin biopsies may be done as a source of germline DNA.
  Other Names: Biopsy

SUMMARY:
The development of next generation sequencing (NGS) techniques, including whole genome (WGS), exome (WES) and RNA sequencing has revolutionized the ability of investigators to query the molecular mechanisms underlying tumor formation. Through the Pediatric Cancer Genome Project (PCGP), investigators at St. Jude Children's Research Hospital (SJCRH) have successfully used NGS approaches to evaluate more than 1,000 pediatric cancers ranging from hematologic malignancies to central nervous system (CNS) and non-CNS solid tumors. From these and related studies, it has become clear that genomic approaches can accurately classify tumors into distinct pathologic and prognostic subtypes and detect alterations in cellular pathways that may serve as novel therapeutic targets. Collectively, these studies suggest that by characterizing the genomic make-up of individual tumors, investigators will be able to develop personalized and potentially more effective cancer treatments and/or preventive measures.

This protocol was initially enacted to usher NGS approaches into routine clinical care. During the initial phase of the G4K protocol, 310 participants were recruited and enrolled onto the study. Tumor and/or germline sequencing was completed on all 310 patients, with 253 somatic reports generated (representing 96% of the 263 participants for whom tumor tissue was available and analyzed) and 301 germline reports generated (100% of the 301 participants who agreed to the receipt of germline results). Analyses of the study data are ongoing with plans to prepare initial manuscripts within the next several months. Due to the successful initial execution of the G4K protocol, clinical genomic sequencing of tumor and germline samples is now offered as part of standard clinical care for pediatric oncology patients at St. Jude.

The G4K protocol has now been revised. With the revision, the study team will record, store and analyze germline and tumor genomic information. Through the collection of these data, we will examine how germline mutations in 150 cancer predisposition genes influence clinical presentation, tumor histology, tumor genomic findings, response to therapy and long-term outcomes. The overall goals of this research are to further define the prevalence, spectrum and heritability of germline variants in these genes and to decipher how germline mutations influence the phenotypes of an expanding array of cancer predisposition syndromes. These studies allow us to provide more accurate genetic counseling and management strategies to future children harboring mutations in these genes.

This remains a non-therapeutic study. Investigators anticipate a sample size of approximately 2500 patients who will be recruited over the next 7 years.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To use clinical genomic sequencing to define the prevalence and spectrum of germline mutations in cancer predisposition genes in children with cancer.
* For those identified with germline mutations, to correlate germline genomic information with clinical presentation, tumor genomic findings, treatment response, and outcome.

OTHER PRESPECIFIED OBJECTIVES:

* To generate and analyze data describing patient/parent perceptions of genomic investigations and research at various time points throughout the study.
* To generate and analyze data surrounding the return of genomic sequencing results, examine patient/parent understanding of these results and assess the impact of results on patients and families.
* To determine the feasibility and reliability of performing WES and RNA sequencing on derivatives from formalin-fixed, paraffin-embedded (FFPE) tumor samples alongside the analysis of matched frozen tumor and germline samples.

For participants who give consent, a normal tissue sample will be obtained and used for WGS, WES and RNA sequence analysis. A defined list of 150 genes will be analyzed for reporting using the normal tissue. Once the results of these analyses are available, they will be disclosed to physicians, patients and parents. Mixed measures approaches will be used to assess understanding, acceptance and impact of genomic results on patients and parents. During the course of the study, the investigators anticipate the list of genes to be reported using normal tissue to change due to advances in the literature or other evidence linking additional genes to tumor formation and cancer risk, and new lists may be defined.

To assess provider, patient and family understanding and describe the impacts of genomic testing and return of results, this study will also incorporate administration of surveys and semi-structured interviews. Surveys and interviews are optional, but will be offered to all primary SJCRH providers, as well as all eligible participants and parents, regardless of whether or not they consent to pursue the genomic testing.

A sample of blood or a skin biopsy will be obtained as a source of germline DNA. This sample is necessary as it is the comparator against which tumor samples are evaluated. Skin biopsies may be done on patients who have a diagnosis where peripheral blood is likely to be contaminated by tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* St. Jude patients prospectively identified at the time of study activation with a diagnosed solid or liquid tumor (benign or malignant).
* Adequate tissue must be available (e.g. sufficient germline and/or tumor tissue, from which >1 µg DNA and >0.1 µg RNA must be isolated). Patients who have no tumor tissue available may enroll using only germline sample.

Exclusion Criteria:

* Past history of hematopoietic stem cell transplantation (or other condition that would result in hematopoietic cell DNA failing to match host tissue DNA).
* Tumor or germline tissue not meeting the criteria listed above.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Participants who are unable to read, write or converse fluently in English or Spanish will be excluded from Prespecified Objectives 3 and 4.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be patients at St. Jude Children's Research Hospital (SJCRH) with diagnoses of hematological, solid or central nervous system tumors who agree to participate in this study and their parents or legally authorized representatives who consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-08-28 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall success rate | Approximately 3 months after study enrollment
  Success is defined by the combined successes of (1) quality interpretable genomic data are generated from sequencing tumor and germline tissues, and (2) communicating genomic test results to the primary SJCRH oncologist and the patient and his/her parents.
  The Binomial proportion of successful performance will be estimated by the sample proportion and the 99% confidence interval based on the normal approximation. Sample size is 400.
Number and type of somatic genetic variants and germline genetic variants | Approximately 3-4 months after the germline sample is obtained
  WGS, WES and RNA sequence data will be used to identify and characterize somatic genetic variants of pathological significance and germline genetic variants associated with increased cancer risk. Descriptive statistics, such as counts and proportions of variants associated with increased cancer risk will be computed within each patient and in each disease type.

OTHER OUTCOMES:
Proportion of parents/participants by perception of genomic testing | At study end (up to 13 months after last participant enrollment)
  Parent/participant perceptions of genomic investigations and research will be assessed using audiotaped conversations and surveys. Results will be summarized by descriptive statistics.
Number of participants/parents by level of understanding | At study end (up to 13 months after last participant enrollment)
  Research participant/parent understanding of genomic results and the impact of results on research participants and their families will be assessed by analysis of audiotaped conversations and survey results. Results will be summarized by descriptive statistics
Proportion of successful sequences of formalin-fixed, paraffin-embedded (FFPE) samples | Approximately 3 months after enrollment
  To assess the practicability, proportions of FFPE samples that can be successfully sequenced will be estimated along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Kim E. Nichols, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Johnson LM, Mandrell BN, Li C, Lu Z, Gattuso J, Harrison LW, Mori M, Ouma AA, Pritchard M, Sharp KMH, Nichols KE. Managing Pandora's Box: Familial Expectations around the Return of (Future) Germline Results. AJOB Empir Bioeth. 2022 Jul-Sep;13(3):152-165. doi: 10.1080/23294515.2022.2063994. Epub 2022 Apr 26. PMID 35471132
- [Derived] Maciaszek JL, Oak N, Chen W, Hamilton KV, McGee RB, Nuccio R, Mostafavi R, Hines-Dowell S, Harrison L, Taylor L, Gerhardt EL, Ouma A, Edmonson MN, Patel A, Nakitandwe J, Pappo AS, Azzato EM, Shurtleff SA, Ellison DW, Downing JR, Hudson MM, Robison LL, Santana V, Newman S, Zhang J, Wang Z, Wu G, Nichols KE, Kesserwan CA. Enrichment of heterozygous germline RECQL4 loss-of-function variants in pediatric osteosarcoma. Cold Spring Harb Mol Case Stud. 2019 Oct 23;5(5):a004218. doi: 10.1101/mcs.a004218. Print 2019 Oct. PMID 31604778
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols